CLINICAL TRIAL: NCT02420704
Title: Effect of Endometrial Thickness on IVF Outcome: a Prospective Observational Study of Both Cleavage Stage and Blastocyst Stage Embryo Transfer Cycles
Brief Title: Effect of Endometrial Thickness on IVF Outcome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Yingpu Sun, Director of Reproductive Medical Center, The First Affiliated Hospital of Zhengzhou University
Other Study IDs: RMCZZU-Endometrial thickness
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Infertility
Keywords: IVF; endometrial thickness; cleavage stage embryo; blastocyst stage embryo; Ongoing pregnancy rate
MeSH Terms: conditions — Infertility | interventions — Embryo Transfer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- Cleavage stage-thin endometrial: Patients transferred with cleavage stage embryo, with endometrial thickness ≤7mm on the day of HCG (human chorionic gonadotropin) administration for fresh cycles, or on the day starting to use progesterone for frozen thawed cycles.
  Interventions: Procedure: Embryo transfer
- Cleavage stage-medium endometrial: Patients transferred with cleavage stage embryo, with endometrial thickness 8-13mm on the day of HCG (human chorionic gonadotropin) administration for fresh cycles, or on the day starting to use progesterone for frozen thawed cycles.
  Interventions: Procedure: Embryo transfer
- Cleavage stage-thick endometrial: Patients transferred with cleavage stage embryo, with endometrial thickness ≥14mm on the day of HCG (human chorionic gonadotropin) administration for fresh cycles, or on the day starting to use progesterone for frozen thawed cycles.
  Interventions: Procedure: Embryo transfer
- Blastocyst stage-thin endometrial: Patients transferred with blastocyst stage embryo, with endometrial thickness ≤7mm on the day of HCG (human chorionic gonadotropin) administration for fresh cycles, or on the day starting to use progesterone for frozen thawed cycles.
  Interventions: Procedure: Embryo transfer
- Blastocyst stage-medium endometrial: Patients transferred with blastocyst stage embryo, with endometrial thickness 8-13mm on the day of HCG (human chorionic gonadotropin) administration for fresh cycles, or on the day starting to use progesterone for frozen thawed cycles.
  Interventions: Procedure: Embryo transfer
- Blastocyst stage-thick endometrial: Patients transferred with blastocyst stage embryo, with endometrial thickness ≥14mm on the day of HCG (human chorionic gonadotropin) administration for fresh cycles, or on the day starting to use progesterone for frozen thawed cycles.
  Interventions: Procedure: Embryo transfer

INTERVENTIONS:
Procedure: Embryo transfer — For fresh cycles, embryos were transferred 3-5 days after oocyte retrieval; For frozen thawed cycles, embryos were transferred 3-5 days after starting to use progesterone based on the stage of cryopreservation.

SUMMARY:
Although many studies have evaluated the relationship between endometrial thickness and IVF outcome, the results are still controversial. We notice that, during our daily work, for patients undergoing cleavage stage embryo transfer, endometrial thickness seems to have a huge impact on IVF outcome; however, for blastocyst stage embryo transfers, IVF outcome seems to have little association with endometrial thickness. Thus, the aim of this prospective observational study is to explore the relationship between endometrial thickness and IVF outcome in patients undergoing cleavage stage and blastocyst stage embryo transfers, respectively.

ELIGIBILITY:
Inclusion Criteria:

* age between 22-38 years old;
* the first cycle of IVF treatment with standard long protocol;
* transfrred with at least two high quality cleavage stage embryos, or with at least one high quality blastocyst stage embryo.

Exclusion Criteria:

* PGD cycles;
* gamete donation cycles

Ages: 22 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients transfrred with at least two high quality cleavage stage embryos, or with at least one high quality blastocyst stage embryo.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 12 weeks after embryo transfer
  An ongoing pregnancy was defined as a pregnancy with a positive heartbeat by ultrasound after 12 weeks gestation.

CONTACTS AND LOCATIONS:
Overall Officials: Yingpu Sun, M.D, Principal Investigator — Reproductive Medical Centre
Locations (1):
- Reproductive Medical Center, First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

REFERENCES:
- [Background] Wu Y, Gao X, Lu X, Xi J, Jiang S, Sun Y, Xi X. Endometrial thickness affects the outcome of in vitro fertilization and embryo transfer in normal responders after GnRH antagonist administration. Reprod Biol Endocrinol. 2014 Oct 9;12:96. doi: 10.1186/1477-7827-12-96. PMID 25296555
- [Background] Zhao J, Zhang Q, Wang Y, Li Y. Endometrial pattern, thickness and growth in predicting pregnancy outcome following 3319 IVF cycle. Reprod Biomed Online. 2014 Sep;29(3):291-8. doi: 10.1016/j.rbmo.2014.05.011. Epub 2014 Jun 13. PMID 25070912
- [Background] Kasius A, Smit JG, Torrance HL, Eijkemans MJ, Mol BW, Opmeer BC, Broekmans FJ. Endometrial thickness and pregnancy rates after IVF: a systematic review and meta-analysis. Hum Reprod Update. 2014 Jul-Aug;20(4):530-41. doi: 10.1093/humupd/dmu011. Epub 2014 Mar 23. PMID 24664156